CLINICAL TRIAL: NCT05788029
Title: Comparing Laparoscopic and Open Pancreaticoduodenectomy for Nonpancreatic Periampullary Adenocarcinomas
Acronym: NPPC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Fudan University (Other); The First Affiliated Hospital of Dalian Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The Third Affiliated Hospital of Soochow University (Other); Shanxi Province Cancer Hospital (Other); Army Medical University, China (Other); Qilu Hospital of Shandong University (Other); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of University of South China (Other); First Affiliated Hospital of Harbin Medical University (Other); Chongqing General Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Prof, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJDBPS14; TJDBPS14 (Other: Tongji Hospital)
Record Dates: First submitted 2022-11-30; First posted 2023-03-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-03

CONDITIONS: Periampullary Adenocarcinoma
Keywords: non-pancreatic periampullary adenocarcinoma; laparoscopic pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laparoscopic pancreaticoduodenectomy (Experimental): laparoscopic pancreaticoduodenectomy
  Interventions: Procedure: laparoscopic pancreaticoduodenectomy
- open pancreaticoduodenectomy (Active Comparator): open pancreaticoduodenectomy
  Interventions: Procedure: open pancreaticoduodenectomy

INTERVENTIONS:
Procedure: laparoscopic pancreaticoduodenectomy — laparoscopic pancreaticoduodenectomy
  Arms: laparoscopic pancreaticoduodenectomy
Procedure: open pancreaticoduodenectomy — open pancreaticoduodenectomy
  Arms: open pancreaticoduodenectomy

SUMMARY:
The aim of this study was to evaluate the outcomes of LPD versus OPD in non-pancreatic periampullary adenocarcinoma

DETAILED DESCRIPTION:
The aim of this study was to evaluate the outcomes of LPD versus OPD in non-pancreatic periampullary adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years and 75 years.
2. Histologically confirmed NPPC or clinically diagnosed NPPC by an MDT without histopathologic evidence.
3. Patients feasible to undergo both LPD and OPD ac- cording to MDT evaluations.
4. Patients understanding and willing to comply with this trial.
5. Provision of written informed consent before patient registration.
6. Patients meeting the curative treatment intent in ac- cordance with clinical guidelines.

Exclusion Criteria:

1. Patients with distant metastases, including peritone- al, liver, distant lymph node metastases and involve- ment of other organs.
2. Patients requiring left, central or total pancreatecto- my or other palliative surgery.
3. Preoperative American Society of Anaesthesiologists (ASA) score ≥4.
4. History of other malignant disease
5. Pregnant or breastfeeding women.
6. Patients with serious mental disorders
7. Patients treated with neoadjuvant therapy.
8. Patients with vascular invasion and requiring vascular resection as evaluated by the MDT team according to abdominal imaging data.
9. Body mass index >35 kg/m 2 .
10. Patients participating in any other clinical trials with- in 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
length of hospital stay | 90 days
  defined as the number of nights spent in the hospital from the end of the surgical procedure until discharge or death

SECONDARY OUTCOMES:
1 year OS | 1 year
  1 year OS
mortality | 90 days
  mortality
morbidity | 90 days
  morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Renyi Qin, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Biliary and Pancreatic Surgery, Tongji Hospital, Affiliated Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Share only when contact to Principal Investigator